CLINICAL TRIAL: NCT07354529
Title: Evaluation of Benefits of Date Fruit in the First Trimester of Pregnancy
Brief Title: Date Fruit Benefits to Treat Morning Sickness in First Trimester of Pregnancy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Major Gen (R) Prof Dr Shehla M Baqai, Principal Bahria University Medical College (BUMC) , Bahria University Health Sciences Campus Karachi, Bahria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUHS-IRB#163/25
Record Dates: First submitted 2025-12-18; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy
Keywords: Pregnancy; Dates; Vomiting; Haemoglobin; Morning Sickness of pregnancy; Hyperemesis gravidarum
MeSH Terms: conditions — Vomiting; Hyperemesis Gravidarum | interventions — Chronology as Topic; doxylamine succinate; Vitamin B 6; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Date fruit (Active Comparator): 3 Dates after breakfast
  Interventions: Other: Date fruit
- Antiemetic medication (Active Comparator): Doxylamine succinate 10 mg + Pyridoxine HCl 10 mg
  Interventions: Drug: Doxylamine succinate 10 mg + Pyridoxine HCl 10 mg
- Appropriate Diet only (Active Comparator): Avoidance of high fat foods and enhanced intake of hydrating fruits and vegetables
  Interventions: Other: Diet

INTERVENTIONS:
Other: Date fruit — 3 Dates after breakfast
  Other Names: Date intake in morning
  Arms: Date fruit
Drug: Doxylamine succinate 10 mg + Pyridoxine HCl 10 mg — Doxylamine succinate 10 mg + Pyridoxine HCl 10 mg , One per day
  Other Names: Antiemetic once per day
  Arms: Antiemetic medication
Other: Diet — Avoidance of high in fat foods and enhanced intake of hydrating fruits and vegetables
  Other Names: Diet as per advice
  Arms: Appropriate Diet only

SUMMARY:
The goal of this randomized clinical trial is to evaluate role of date fruit in alleviating morning sickness of pregnancy in pregnant females. The main question[s] it aims to answer [is/are]:

The goal of this randomized clinical trial is to evaluate role of date fruit in

The goal of this randomized clinical trial is to evaluate role of date fruit in alleviating vomiting due to morning sickness of pregnancy and in improving maternal hemoglobin in pregnant females. The main question[s] it aims to answer [are]:

* Role of date fruit in alleviating severity and frequency of vomiting due to morning sickness of pregnancy in pregnant females.
* Role of date fruit in improving haemoglobin levels in pregnant females.
* To assess improvement of severity and frequency of vomiting due to morning sickness of pregnancy and improvement of hemoglobin levels in pregnant females, researchers will compare date fruit intake with antiemetic medication doxylamine succinate 10 mg + pyridoxine HCl 10 and diet only.

DETAILED DESCRIPTION:
A randomized Controlled trial to assess benefits of date fruit in morning sickness of pregnancy symptoms, inclusive of nausea and vomiting and to improve haemoglobin levels in pregnant females.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females in 18 to 45 year old age group

Exclusion Criteria:

1. Females in 18 to 45 year old age group who are not pregnant.
2. Females less than 18 years old.
3. Females over 45 years.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females only
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 12 Weeks
  Complete blood picture (Laboratory diagnostic tests)
Vomiting | 12 Weeks
  PUQE-24 Score Unabbreviated scale title : The Pregnancy-Unique Quantification of Emesis and Nausea (PUQE-24) Minimum Value : 4-6 (Mild) Maximum Value : ≥13 (Severe) Higher Scores mean worst outcome

SECONDARY OUTCOMES:
Fatigue level | 12 weeks
  FAS Unabbreviated scale title: Fatigue Assessment Scale (FAS)
  Minimum Value : Less less than 22 Maximum Value : 35 or more indicates severe fatigue Higher Scores mean worst outcome
Dietary Recall | 12 weeks
  Direct compliance inquired via telephonic communication on regular basis

CONTACTS AND LOCATIONS:
Overall Officials: Shehla M Baqai, MBBS, FCPS, FICS, Principal Investigator — Bahria University Health Sciences Campus Karachi
Locations (1):
- PNS SHIFA Hospital , Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No